CLINICAL TRIAL: NCT00000492
Title: Beta-Blocker Heart Attack Trial (BHAT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 11
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 1981-10

CONDITIONS: Arrhythmia; Cardiovascular Diseases; Coronary Disease; Death, Sudden, Cardiac; Heart Diseases; Myocardial Infarction; Myocardial Ischemia; Ventricular Fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Cardiovascular Diseases; Coronary Disease; Death, Sudden, Cardiac; Heart Diseases; Myocardial Infarction; Myocardial Ischemia; Ventricular Fibrillation | interventions — Propranolol

INTERVENTIONS:
Drug: propranolol

SUMMARY:
To determine whether the regular administration of the beta-blocker drug propranolol to people who had had at least one documented myocardial infarction would result in a significant reduction of mortality from all causes over the follow-up period. Eligible volunteer patients were recruited to participate in a double-blind clinical trial within 21 days after the onset of the acute event. One-half of the patients were randomly assigned to a beta-blocking drug (propranolol) and one-half to a placebo. The trial also evaluated the effect of propranolol on incidences of coronary heart disease mortality, sudden cardiac death, and nonfatal myocardial infarction plus coronary heart disease mortality in persons with documented previous myocardial infarction.

DETAILED DESCRIPTION:
BACKGROUND:

Survivors of a documented myocardial infarction are recognized as having a high risk of dying relative to the general population. Serious arrhythmias, occurring with or without evidence of new infarction, are a common cause of death in this population. Theoretically, an agent which (1) can block the sympathetic nervous activity thought to be involved in precipitating sudden death and (2) has non-neurogenic antiarrhythmic properties would be of value to people with coronary heart disease. Propranolol, like other beta- blocking agents, has these as well as other properties and therefore might be expected to prevent or retard complications of coronary heart disease such as serious arrhythmias. This would be reflected in a decrease in mortality due to coronary heart disease.

A workshop on chronic antiarrhythmic therapy reviewed contemporary experimental data and clinical practice and recommended that a clinical trial be undertaken to clearly show the effects of beta-blocking drugs on mortality. Subsequently, such a trial was approved by the Clinical Applications and Prevention Advisory Committee, by the Cardiology Advisory Committee, and by the National Heart, Lung, and Blood Advisory Council.

The study protocol was reviewed in February 1978 and recommended for approval by the policy-data monitoring board and ad hoc members. The protocol was approved by the Director of NHLBI in March 1978. Recruitment started on June 19, 1978, and ended in October 1980. A total of 3,837 patients were randomized. Units which participated in the trial included 32 clinical centers, an EKG center, a central laboratory, a coordinating center, a 1-hour ambulatory ECG center, a 24-hour ambulatory EKG center, and an EKG tape quality control center.

DESIGN NARRATIVE:

A randomized, double-blind design with single experimental and control groups. Patients were recruited while in the hospital for an acute myocardial infarction and were enrolled in the study before discharge. Eligible patients fulfilled the study definition of an acute myocardial infarction. The diagnosis was based either on electrocardiographic records showing evolving QRS segment changes or on ST segment and T wave changes together with enzyme changes and appropriate clinical history. One-half of the patients were placed on therapy using a beta-blocking drug (propranolol). The other half received a placebo. The prescribed maintenance dosage of propranolol was either l80 or 240 mgs/day, depending upon serum drug levels. Intervention duration averaged 25 months.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
Men and women, ages 30 to 69. Documented myocardial infarction.

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1977-09; Study Completion 1981-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Barker — Salt Lake Clinic Research Foundation; Nemat Borhani — University of California, Davis; Gerald Breneman — Henry Ford Hospital; Frank Canosa — Miami Heart Institute; Robert Capone — Rhode Island Hospital; Richard Crow — University of Minnesota; Alan Forker (participated until Feb — University of Nebraska; Peter Gazes — University of South Carolina; John Gregory — Atlantic Health System; John Grover — Kaiser Foundation Research Institute; Olga Haring — Northwestern University; Julian Haywood — University of Southern California; William Holmes — Lankenau Hospital; Frank Ibbott — Bio-Science Laboratories; Robert Kohn — State University of New York; Robert Kramer — Long Island Jewish-Hillside Medical Center; Peter Kuo — New Jersey College of Medicine and Dentistry-Rutgers; Charles Laubach — Geisinger Clinic; Edgar Lichstein — Maimonides Medical Center; Louis Matthews — Dartmouth-Hitchcock Medical Center; Gordon Maurice — Providence Medical Center; J. McNamara — Pacific Health Research Institute; E. Michau — Veterans Administration Hospital; Richard Miller — Baylor College of Medicine; Joel Morganroth — Anthropometrics Heart Clinic; Marvin Murphy; Robert Peters — University of California; Thaddeus Prout — Greater Baltimore Medical Center; Phillip Ranheim — MOUNT SINAI HOSPITAL; David Richardson — Medical College of Virginia; Robert Schlant — Emory University; James Schoenberger — Rush-Presbyterian-St.Luke's Hospital; Pierre Theroux — Montreal Heart Institute; Pantel Vokonas — Boston University; James Walsh — Veterans Administration Hospital; Gary Wilner — Endeavor Health; Paul Yu — University of Rochester

REFERENCES:
- [Background] Beta-Blocker Heart Attack Trial Study Group: Beta-Blocker Heart Attack Trial Study Protocol. DHHS Pub. No. (NIH)81-2209, 1980.
- [Background] The beta-blocker heart attack trial. beta-Blocker Heart Attack Study Group. JAMA. 1981 Nov 6;246(18):2073-4. PMID 7026815
- [Background] Howard JM, DeMets D. How informed is informed consent? The BHAT experience. Control Clin Trials. 1981 Dec;2(4):287-303. doi: 10.1016/0197-2456(81)90019-2. PMID 6120794
- [Background] Beta Blocker Heart Attack Trial: design features. Control Clin Trials. 1981 Dec;2(4):275-85. doi: 10.1016/0197-2456(81)90018-0. PMID 6120793
- [Background] A randomized trial of propranolol in patients with acute myocardial infarction. I. Mortality results. JAMA. 1982 Mar 26;247(12):1707-14. doi: 10.1001/jama.1982.03320370021023. PMID 7038157
- [Background] Furberg CD, Byington RP. What do subgroup analyses reveal about differential response to beta-blocker therapy? The Beta-Blocker Heart Attack Trial experience. Circulation. 1983 Jun;67(6 Pt 2):I98-101. PMID 6133654
- [Background] A randomized trial of propranolol in patients with acute myocardial infarction. II. Morbidity results. JAMA. 1983 Nov 25;250(20):2814-9. doi: 10.1001/jama.1983.03340200048027. PMID 6358542
- [Background] Goldstein S. The Beta-Blocker Heart Attack Trial in perspective. Cardiology. 1983;70(5):255-62. doi: 10.1159/000173602. PMID 6141847
- [Background] Shulman RS, Herbert PN, Capone RJ, McClure D, Hawkins CM, Henderson LO, Saritelli A, Campbell J. Effects of propranolol on blood lipids and lipoproteins in myocardial infarction. Circulation. 1983 Jun;67(6 Pt 2):I19-21. PMID 6851036
- [Background] Lichstein E, Morganroth J, Harrist R, Hubble E. Effect of propranolol on ventricular arrhythmia. The beta-blocker heart attack trial experience. Circulation. 1983 Jun;67(6 Pt 2):I5-10. PMID 6342839
- [Background] Goldstein S. Propranolol therapy in patients with acute myocardial infarction: the Beta-Blocker Heart Attack Trial. Circulation. 1983 Jun;67(6 Pt 2):I53-7. PMID 6342840
- [Background] Byington RP. Beta-blocker heart attack trial: design, methods, and baseline results. Beta-blocker heart attack trial research group. Control Clin Trials. 1984 Dec;5(4):382-437. doi: 10.1016/s0197-2456(84)80017-3. PMID 6151483
- [Background] Haywood LJ. Coronary heart disease mortality/morbidity and risk in blacks. I: Clinical manifestations and diagnostic criteria: the experience with the Beta Blocker Heart Attack Trial. Am Heart J. 1984 Sep;108(3 Pt 2):787-93. doi: 10.1016/0002-8703(84)90672-0. PMID 6148005
- [Background] Furberg CD, Hawkins CM, Lichstein E. Effect of propranolol in postinfarction patients with mechanical or electrical complications. Circulation. 1984 Apr;69(4):761-5. doi: 10.1161/01.cir.69.4.761. PMID 6365352
- [Background] DeMets DL, Hardy R, Friedman LM, Lan KK. Statistical aspects of early termination in the beta-blocker heart attack trial. Control Clin Trials. 1984 Dec;5(4):362-72. doi: 10.1016/s0197-2456(84)80015-x. PMID 6151482
- [Background] Byington RP, Curb JD, Mattson ME. Assessment of double-blindness at the conclusion of the beta-Blocker Heart Attack Trial. JAMA. 1985 Mar 22-29;253(12):1733-6. PMID 3974051
- [Background] Byington R, Goldstein S. Association of digitalis therapy with mortality in survivors of acute myocardial infarction: observations in the Beta-Blocker Heart Attack Trial. J Am Coll Cardiol. 1985 Nov;6(5):976-82. doi: 10.1016/s0735-1097(85)80297-7. PMID 4045047
- [Background] Morganroth J, Lichstein E, Byington R. Beta-Blocker Heart Attack Trial: impact of propranolol therapy on ventricular arrhythmias. Prev Med. 1985 May;14(3):346-57. doi: 10.1016/0091-7435(85)90061-1. PMID 3903736
- [Background] Bell RL, Curb JD, Friedman LM, McIntyre KM, Payton-Ross C. Enhancement of visit adherence in the national beta-blocker heart attack trial. Control Clin Trials. 1985 Jun;6(2):89-101. doi: 10.1016/0197-2456(85)90114-x. PMID 3891227
- [Background] Bell RL, Curb JD, Friedman LM, Payne GH. Termination of clinical trials: the beta-blocker heart attack trial and the hypertension detection and follow-up program experience. Control Clin Trials. 1985 Jun;6(2):102-11. doi: 10.1016/0197-2456(85)90115-1. PMID 4006483
- [Background] Walle T, Byington RP, Furberg CD, McIntyre KM, Vokonas PS. Biologic determinants of propranolol disposition: results from 1308 patients in the Beta-Blocker Heart Attack Trial. Clin Pharmacol Ther. 1985 Nov;38(5):509-18. doi: 10.1038/clpt.1985.216. PMID 4053488
- [Background] Goldstein S, Byington R. The Beta Blocker Heart Attack Trial: recruitment experience. Control Clin Trials. 1987 Dec;8(4 Suppl):79S-85S. doi: 10.1016/0197-2456(87)90010-9. PMID 2894282
- [Background] Furberg CD, Friedman LM, MacMahon SW: Women as Participants in Trials of the Primary and Secondary Prevention of Cardiovascular Disease: Part II. Secondary Prevention: The Beta-Blocker Heart Attack Trial and the Aspirin Myocardial Infarction Study, in: Coronary Heart Disease in Women. Ed Eaker, B Packard, NK Wenger, TB Clarkson, HA Tyroler (Eds). New York, Haymarket Doyma, pp 241-246, 1987.
- [Background] Kostis JB, Byington R, Friedman LM, Goldstein S, Furberg C. Prognostic significance of ventricular ectopic activity in survivors of acute myocardial infarction. J Am Coll Cardiol. 1987 Aug;10(2):231-42. doi: 10.1016/s0735-1097(87)80001-3. PMID 2439559
- [Background] Peters RW, Byington R, Arensberg D, Friedman LM, Romhilt DW, Barker A, Laubach C, Wilner GW, Goldstein S. Mortality in the beta blocker heart attack trial: circumstances surrounding death. J Chronic Dis. 1987;40(1):75-82. doi: 10.1016/0021-9681(87)90098-1. PMID 3543049
- [Background] Davis BR, Furberg CD, Williams CB. Survival analysis of adverse effects data in the Beta-Blocker Heart Attack Trial. Clin Pharmacol Ther. 1987 Jun;41(6):611-5. doi: 10.1038/clpt.1987.83. PMID 3555942
- [Background] Davis BR, Friedman LM, Lichstein E. Are 24 hours of ambulatory ECG monitoring necessary for a patient after infarction? Am Heart J. 1988 Jan;115(1 Pt 1):83-91. doi: 10.1016/0002-8703(88)90521-2. PMID 3276112
- [Background] Peters RW, Muller JE, Goldstein S, Byington R, Friedman LM. Propranolol and the morning increase in the frequency of sudden cardiac death (BHAT Study). Am J Cardiol. 1989 Jun 15;63(20):1518-20. doi: 10.1016/0002-9149(89)90019-2. No abstract available. PMID 2729140
- [Background] Peters RW, Byington RP, Barker A, Yusuf S. Prognostic value of prolonged ventricular repolarization following myocardial infarction: the BHAT experience. The BHAT Study Group. J Clin Epidemiol. 1990;43(2):167-72. doi: 10.1016/0895-4356(90)90180-w. PMID 2406377
- [Background] Byington RP, Worthy J, Craven T, Furberg CD. Propranolol-induced lipid changes and their prognostic significance after a myocardial infarction: the Beta-Blocker Heart Attack Trial experience. Am J Cardiol. 1990 Jun 1;65(20):1287-91. doi: 10.1016/0002-9149(90)91314-v. PMID 2188492
- [Background] Gheorghiade M, Schultz L, Tilley B, Kao W, Goldstein S. Effects of propranolol in non-Q-wave acute myocardial infarction in the beta blocker heart attack trial. Am J Cardiol. 1990 Jul 15;66(2):129-33. doi: 10.1016/0002-9149(90)90575-l. PMID 2196771
- [Background] Peters RW. Propranolol and the morning increase in sudden cardiac death: (the beta-blocker heart attack trial experience). Am J Cardiol. 1990 Nov 6;66(16):57G-59G. doi: 10.1016/0002-9149(90)90398-k. PMID 2239715
- [Background] Gheorghiade M, Schultz L, Tilley B, Kao W, Goldstein S. Natural history of the first non-Q wave myocardial infarction in the placebo arm of the Beta-Blocker Heart Attack Trial. Am Heart J. 1991 Dec;122(6):1548-53. doi: 10.1016/0002-8703(91)90270-r. PMID 1957749
- [Background] Gheorghiade M, Shivkumar K, Schultz L, Jafri S, Tilley B, Goldstein S. Prognostic significance of electrocardiographic persistent ST depression in patients with their first myocardial infarction in the placebo arm of the Beta-Blocker Heart Attack Trial. Am Heart J. 1993 Aug;126(2):271-8. doi: 10.1016/0002-8703(93)91039-h. PMID 8337995
- [Background] Friedman LM, Byington RP. Assessment of angina pectoris after myocardial infarction: comparison of "Rose Questionnaire" with physician judgment in the Beta-Blocker Heart Attack Trial. Am J Epidemiol. 1985 Apr;121(4):555-62. doi: 10.1093/oxfordjournals.aje.a114033. PMID 3893101
- [Background] Furberg C. The beta-blocker heart attack trial. Br J Clin Pharmacol. 1982;14 Suppl 1(Suppl 1):3S-5S. doi: 10.1111/j.1365-2125.1982.tb02053.x. No abstract available. PMID 6126206
- [Background] Hawkins CM, Richardson DW, Vokonas PS. Effect of propranolol in reducing mortality in older myocardial infarction patients. The Beta-Blocker Heart Attack Trial experience. Circulation. 1983 Jun;67(6 Pt 2):I94-7. PMID 6342843
- [Background] Friedman LM, Byington RP, Capone RJ, Furberg CD, Goldstein S, Lichstein E. Effect of propranolol in patients with myocardial infarction and ventricular arrhythmia. J Am Coll Cardiol. 1986 Jan;7(1):1-8. doi: 10.1016/s0735-1097(86)80250-9. PMID 3510232
- Available data/document: Individual Participant Data Set: BHAT — http://biolincc.nhlbi.nih.gov/studies/bhat/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/bhat/